CLINICAL TRIAL: NCT02610595
Title: A Prospective, Multi-center Study of the Chinese Medicine for the Treatment of MDR Membranous Nephropathy in the Traditional Chinese Medicine (a Herbal Formula for Invigorating Spleen and Benefiting qi and Promoting Blood Circulation)
Brief Title: Study on the Therapeutic Effect of TCM Treatment for MDR MN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Fudan University (Other); Ruijin Hospital (Other); Shanghai 6th People's Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Changhai Hospital (Other); Shanghai Putuo District Center Hospital (Other); ShuGuang Hospital (Other); Shanghai Yueyang Integrated Medicine Hospital (Other); Shanghai Changzheng Hospital (Other); Shanghai Minhang Central Hospital (Other); Zhujiang Hospital (Other); Guangxi Traditional Chinese Medical University (Other); Huashan Hospital (Other); The First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine (Other); Xinqiao Hospital of Chongqing (Other); Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other); Nanjing University of Traditional Chinese Medicine (Other); Tongji Hospital (Other); Chinese Academy of Sciences (Other Government); RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZY3-CCCX-3-2001
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-08

CONDITIONS: Idiopathic Membranous Nephropathy
Keywords: Idiopathic Membranous Nephropathy; Jianpiyiqi Recipe; Huoxuejiedu Recipe; Effectiveness; Safety
MeSH Terms: conditions — Glomerulonephritis, Membranous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- experimental group (Experimental): Jianpixiaozhong particles and Wuse Dietotherapy
  Interventions: Drug: Jianpixiaozhong particles and Wuse Dietotherapy

INTERVENTIONS:
Drug: Jianpixiaozhong particles and Wuse Dietotherapy — Jianpixiaozhong particles: Three packs once,bid po; Wuse Dietotherapy: one packs once,bid po

SUMMARY:
To evaluate the effectiveness and safety of the Chinese medicine treatment for multiple drug resistance of MN patients with Jianpiyiqi and Huoxuejiedu Recipe.

DETAILED DESCRIPTION:
Based on previous research, the investigators hoping to identity the standard treatment program for MDR IMN patients with high treatment difficulty, TCM syndrome of s Pixushuifan. Subsequently, to evaluate the effectiveness and safety of the Chinese medicine treatment for multiple drug resistance of MN patients with Jianpiyiqi and Huoxuejiedu Recipe. With twenty national-grade III hospital of to formed TCM Comprehensive treatment plan and to evaluate the effectiveness and safety of the Chinese medicine treatment for multiple drug resistance of MN patients with Jianpiyiqi and Huoxuejiedu Recipe. Furthermore, search for potential diagnostic predictor in IMN by Proteomics and Metabolomics. The investigators purpose is improve the clinical remission rate of MN, further establish the treatment of TCM in the treatment of MN.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years;
2. Gender, nationality;
3. Pixushuifan syndrome, IMN confirmed by renal biopsy and clinical examination;
4. Treatment invalided by two or more than two kinds of Hormone or immunosuppressive agents ;
5. CKD phase 1-3（eGFR（EPI Formula）≥30ml/min/1.73m2）

Exclusion Criteria:

1. Progressive MN (progressive renal impairment, renal biopsy confirmed Necrotic Vasculitis and Large crescent formation>50%), combined with IgA nephropathy, diabetic nephropathy and other renal diseases;
2. Anti-nuclear antibodies, double stranded DNA, ANCA or other indicators of immune disorders;
3. Active hepatitis B and liver function test sustained abnormal;
4. Patients with malignant tumor or have a history of cancer, HIV infection, history of mental illness, acute central nervous system diseases, severe gastrointestinal diseases;
5. Merger with other serious disease and dysfunction of the organ;
6. Gravid or lactation woman;
7. Other clinical trials are being studied.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Remission rate of 24 hours urinary protein quantitative | two weeks to three months

SECONDARY OUTCOMES:
Renal function, glomerular filtration rate (EPI formula), Plasma albumin | two weeks to three months
Blood lipid | half a year
Change of TCM Syndrome | two weeks to three months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nephrology,Longhua Hospital, Shanghai, China